CLINICAL TRIAL: NCT03343769
Title: Study of the Relationship Between the Strength of Ankle Movement Muscles and Postural Parameters in Elderly Fallers: Towards New Strategies for Screening and Management
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: GREMEAUX DRCI 2009-2
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Persons Who Have Experienced a Sudden Uncontrolled Fall in the Absence of Outside Factors in the 6 Months Preceding the Consultation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient
  Interventions: Other: BERG scale; Other: Functional tests; Other: Measurement of balance on a force platform; Other: Measurement of maximal moment of the plantar flexor and dorsiflexor muscles; Other: Measurement of the moment of the plantar flexors and dorsiflexors corresponding to RMS activity during balance measurements
- Control
  Interventions: Other: BERG scale; Other: Functional tests; Other: Measurement of balance on a force platform; Other: Measurement of maximal moment of the plantar flexor and dorsiflexor muscles; Other: Measurement of the moment of the plantar flexors and dorsiflexors corresponding to RMS activity during balance measurements

INTERVENTIONS:
Other: BERG scale — Complete the BERG balance scale
Other: Functional tests — timed up and go, Mini motor test, retropulsion test
Other: Measurement of balance on a force platform — 4 trials of 30 seconds x 2 conditions (eyes open; eyes closed)
Other: Measurement of maximal moment of the plantar flexor and dorsiflexor muscles — 5-second repetitions
Other: Measurement of the moment of the plantar flexors and dorsiflexors corresponding to RMS activity during balance measurements — 3 10-second repetitions

SUMMARY:
The quality of life of elderly citizens is to a great extent related to the maintenance of independence. The risk of falling and the loss of autonomy are two frequent problems associated with ageing. Although the impact of falls on functional outcomes and morbi-mortality in the elderly is well-established, the pathophysiological mechanisms underlying these falls are poorly understood. To better assess the risk of falling, numerous studies have investigated the use of dynamic and static posturography. These studies sought to characterise populations of fallers and non-fallers using parameters from postural analysis. Nonetheless, a new concept may emerge: weakening of the ankle movement muscles may be implicated in the age-related deterioration of posture. Even though it has been shown that this decrease occurs earlier and is more severe in fallers, the direct relationship between the strength of ankle movement muscles and balance parameters in elderly fallers has not yet been established. The existence of such a relationship would make it possible on the one hand to facilitate screening for those with a risk of falling, and on the other hand to enrich our understanding of the pathophysiology of the risk of falling. The perspective would therefore be to propose programmes focused on the strengthening of these deficient muscles.

ELIGIBILITY:
Inclusion Criteria:

Control group:

* Subjects who have provided written informed consent
* Subjects with national health insurance cover
* Subjects aged between 60 and 90 years old
* Able to understand simple instructions and exercise instructions and to provide informed consent
* with no diseases that could compromise postural abilities and ankle muscle strength.
* Subjects who have not experience a sudden uncontrolled fall in the absence of outside factors in the 6 months preceding inclusion.

Patients group

* Subjects who have provided written informed consent
* Subjects with national health insurance cover
* Subjects aged between 60 and 90 years old
* Able to understand simple instructions and exercise instructions and to provide informed consent
* Subjects who have experienced at least one sudden uncontrolled fall in the absence of outside factors in the 6 months preceding inclusion.

Exclusion Criteria:

* Acute balance disorders (central vestibular syndrome, infection or toxic cause)
* Chronic vestibular disease with proven clinical repercussions
* Any severe neuro-orthopedic disease impairing balance as well as physiological impairments due to ageing Any chronic neurological disorder (stroke, Parkinson syndrome…)
* Any psychiatric disorder able to compromise participation
* Non-corrected vision disorder
* Cancer or any progressive disease
* Treatment with psychotropic agents able to impair vigilance and posture
* Patients under guardianship
* Patients with an ADL score <3 (total of 6 points), reflecting a clinically obvious high risk of falling

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients followed at the Pôle de rééducation et de réadaptation
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The sum of the moments of strength developed by the plantar flexor and dorsiflexor muscles (i.e. combined moment) in both ankles | Through study completion, an average of 1 month
Mean total displacement of the Centre of Pressure in millimetres during the different stabilometry recordings. | Through study completion, an average of 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Cattagni T, Scaglioni G, Laroche D, Gremeaux V, Martin A. The involvement of ankle muscles in maintaining balance in the upright posture is higher in elderly fallers. Exp Gerontol. 2016 May;77:38-45. doi: 10.1016/j.exger.2016.02.010. Epub 2016 Feb 16. PMID 26899564